CLINICAL TRIAL: NCT02586077
Title: Foot and Ankle Clinic Application for Liposomal Related Anesthetic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-13-12E
Record Dates: First submitted 2015-06-01; First posted 2015-10-26 (Estimated); Results first posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Ankle Arthrodesis; Hindfoot Arthrodesis; Tibitalocalceal Arthrodesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exparel (Experimental): Patients will receive a single shot popliteal block (standard of care) and then undergo their standardized procedure. Patients will then receive 20cc Exparel and 10cc of normal saline at the conclusion of the case.
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Exparel

SUMMARY:
The purpose of this study is to review the use of surgeon applied liposomal release anesthetic (Exparel) for post operative analgesia.

Hypothesis: Surgeon applied use of liposomal related anesthetic provides excellent post operative analgesia. Immediated and 72 hour narcotic use will be significantly impacted by the use of this modality.

ELIGIBILITY:
Inclusion Criteria:

* Any patient scheduled for ankle arthrodesis, a tibiotalocalcaneal arthrodesis, hindfoot arthrodesis including subtalar, double, triple, or isolated talonavicular arthrodesis
* Patients over the age of 18
* The subject is psychosocially, mentally, and physically able to understand and comply with the requirements of the study

Exclusion Criteria:

* < 18 years of age
* Patients with a history of infection
* Patients diagnosed with neuropathy or any form of numbness or loss of feeling in the arms or legs due to damaged nerves
* Patients having surgery on both feet at the same time
* Patients having any other different type of foot and ankle surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02-01; Primary Completion 2016-06-30 (Actual); Study Completion 2016-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Odum, PhD, Study Director — OrthoCarolina Research Institute; Bruce Cohen, MD, Principal Investigator — OrthoCarolina Foot & Ankle Institute
Locations (1):
- OrthoCarolina, PA, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exparel
Started | 36
Completed | 28
Not Completed | 8
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 4
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Patients completing study
Arm/Group | Exparel
Number analyzed (Participants) | 28
Age, Continuous [Mean (Full Range); unit: years] | 55.6 [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Amount of Narcotic Use
Description: Total morphine milligram equivalence dosing of all narcotic pain medications administered between the surgery and the third post-operative day.
Time Frame: Surgery to post operative day 3
Measure: Mean (Full Range); unit: mg
Arm/Group | Exparel
Number analyzed (Participants) | 28
mg | 236.68 [45 to 570]

2. Secondary Outcome: Visual Analog Scale of Pain (0-10)
Description: Visual Analog Scale (VAS) of pain (0-10); with 10 indicating the greatest amount of pain. Post anesthesia care unit admission, post anesthesia care unit discharge, day of surgery, post operative day 1, post operative day 2, post operative day 3
Time Frame: Post anesthesia care unit admission to post operative day 3
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Exparel
Number analyzed (Participants) | 28
units on a scale
  Post anesthesia care unit admission | 0.96 [0 to 10]
  Post anesthesia care unit discharge | 0.86 [0 to 6]
  Day of Surgery | 2.36 [0 to 7]
  Post-Operative Day 1 | 5.04 [1 to 10]
  Post-operative Day 2 | 3.82 [0 to 10]
  Post-operative Day 3 | 4.29 [0 to 9]

3. Secondary Outcome: Anti-emetic Use
Description: Anti-emetic use (as a binary yes/no) between the admission in the post anesthesia care unit through hospital discharge (i.e. if a patient took an anti-emetic at any point duration the time frame the patient was a yes; if the patient did not take an anti-emetic during the time frame the patient was a no).
Time Frame: After surgery through discharge from hospital, usually 72 hours after surgery (on post operative day 3)
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Data across all patients
Arm/Group | Overall
Number analyzed (Participants) | 28
Participants
  No | 19
  Yes | 9

4. Secondary Outcome: Patient Satisfaction Questionnaire Regarding Post Surgical Pain Relief
Description: Measured at hospital discharge (on post operative day 3). Measured on a scale of 1-5, with 5 being the most satisfaction
Time Frame: Measured at hospital discharge (on post operative day 3)
Measure: Count of Participants; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 28
Participants
  1 | 3
  2 | 3
  3 | 4
  4 | 6
  5 | 12

5. Secondary Outcome: Number of Patients With Post-operative Complications
Description: Any complications occurring between the day of surgery and the first scheduled appointment at our clinic after the surgery.
Time Frame: After surgery to the first scheduled clinic visit, usually 14 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 28
Participants
  No | 27
  Yes | 1

ADVERSE EVENTS:
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 1/36
Other Adverse Events (participants affected / at risk) | 1/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=36)
Increased pain (General disorders) | 1 (1) — Increased pain caused admission to floor from PACU.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=36)
superficial cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) — Developed a superficial cellulitis that required antibiotic treatment. There were no secondary surgical procedures necessary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No